CLINICAL TRIAL: NCT07293962
Title: Liquid S-Platelet Rich Fibrin as a Potential Adjunct in Conservative Closed Periodontal Debridement for Periodontitis Stages II-IV: A Randomized, Split-mouth, 3-month Clinical Trial
Brief Title: 3-Month Clinical Trial of Liquid S-PRF in Periodontal Debridement for Periodontitis Stages II-IV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mahsa University (Other)
Responsible Party: Principal Investigator, Wong Hong Zhang, Dr., Mahsa University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RMC/MAR/2024/EC16
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Periodontitis Stage II; Periodontitis Stage III; Periodontitis (Stage 3); Periodontitis; Periodontitis Chronic Localized Slight; Periodontitis Chronic Generalized Moderate; Periodontitis Chronic Generalized Severe; Periodontitis, Adult; Periodontitis, Chronic
Keywords: periodontal treatment; periodontitis; platelet concentrates; platelet-rich fibrin; nonsurgical; clinical trial; periodontal; nonsurgical periodontal debridement; dental scaling; periodontal diseases; periodontal debridement; nonsurgical periodontal treatment
MeSH Terms: conditions — Periodontitis; Chronic Periodontitis; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Prospective split-mouth, single-blind, randomized controlled trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control half of mouth (Placebo Comparator): Normal saline irrigation after root debridement
  Interventions: Procedure: Normal saline irrigation
- Experimental half of mouth (Experimental): Liquid S-PRF irrigation after root debridement
  Interventions: Drug: Platelet rich fibrin

INTERVENTIONS:
Procedure: Normal saline irrigation — Full mouth scaling or professional mechanical plaque removal, air polishing, and root debridement wherever deep pockets are indicated, then normal saline irrigation after root debridement
  Arms: Control half of mouth
Drug: Platelet rich fibrin — Full mouth scaling or professional mechanical plaque removal, air polishing, and root debridement wherever deep pockets are indicated, then liquid S-PRF irrigation after root debridement
  Arms: Experimental half of mouth

SUMMARY:
What is the purpose of this study? This study is to investigate the effect of a processed blood product in healing after treatment for gum disease. In addition to scaling & root debridement (deep cleaning) that is the standard treatment for periodontitis, this study will test the effectiveness of patient's processed blood in improving healing of diseased gums.

What are the procedures to be followed? First, all patients will undergo dental check-up and X-ray imaging for suitability as a participant for the project. For participants who are eligible and included into study, upper & lower jaws models will be made, and each will be given oral care kit & instructions. The next appointment will be given for scaling & root debridement with local numbing agent in one day. Towards the end of the treatment, a small amount (20 mℓ) of blood will be collected and spun to produce liquid platelet-rich fibrin that is then used to flush the treated gum pockets in half of the mouth. For the treated gum pockets in the opposite half of the mouth, sterile salt water (saline) will be used instead for comparison. Then, follow-up appointments are at monthly intervals until 3 months.

Who should enter the study? Symptoms of gum disease include bleeding and/or receding gums, tooth/teeth appearing longer or feeling shaky/loose/weak, formation of large amount of calculus and/or black/empty space between teeth, frequent/recurrent gum swelling/pus, and/or bad breath.

DETAILED DESCRIPTION:
Introduction: We appreciate your participation in the present study. This study is to investigate the effect of a processed blood product in healing after treatment for severe gum disease.

What is the purpose of this study? This study will test the efficacy of a biomaterial made by processing blood drawn from the participant's own arm that may improve healing once inserted into diseased gum pockets. For comparison, the other material used will be saline, which together with scaling & root debridement forms the basic standard of care protocol for the treatment of periodontitis.

What are the procedures to be followed? Clinical examination will be done on all the participants to screen and check for the suitability to be included as a participant for the project. Panoramic X-ray radiograph(s) will be taken to see the bone height underneath the gums. Included participants will be given oral care instructions & kit, and have alginate molds taken of their upper & lower jaws for making a custom guide. The first appointment will be given for scaling & root debridement with local numbing agent in one day. Towards the end of the treatment, 20 mℓ of blood will be collected from a vein in either arm. The blood will be processed to produce a liquid material that will be irrigated into tested gum pockets. For the other tested sites, saline irrigation will be performed instead. Then, appointment are given at monthly interval to review the results of the treatment until 3 months. Follow-up care will then be provided as necessary, outside the scope of this study.

Who should enter the study? Compliant adults with severe gum disease and having at least 20 teeth. What will be the benefits of the study?

1. To you as a subject? The blood-derived biomaterial may improve gum healing compared to natural unassisted process. The involved procedures will be performed free-of-charge worth around RM 500-4000 as a token of appreciation for your participation. Stipend per appointment will be provided for travel expenses.
2. To the investigator? The investigator can evaluate the clinical parameter.

What are the possible drawbacks? Blood-drawing is required.

Will there be complications? For blood drawing, the risks are not limited to but include risk of injuries, bruising, swelling, infection, and allergic reaction.

For scaling, the risks are not limited to but include risk of choking, accidental swallowing, bleeding, injury to adjacent structures, teeth sensitivity, teeth mobility, recession, swelling, fever, infection, and flare-up in between appointments.

For local numbing agent (anesthesia), the risks are not limited to but include risk of bleeding, swelling, choking, accidentally biting own lips, cheeks, &/or tongue, difficulty swallowing &/or breathing, injury to adjacent structures, nerve injury, inability to close eyes, inability to open mouth, and allergic reaction.

For root debridement, the risks are not limited to but include risk of bleeding, injury to adjacent structures, teeth sensitivity, teeth mobility, recession, swelling, fever, infection, and flare-up in between appointments.

ELIGIBILITY:
Inclusion Criteria:

* Have at least 20 teeth,
* American Society of Anesthesiology class I or II
* Periodontitis stages II-IV
* Bilateral sites of deep periodontal pockets ≥5 mm

Exclusion Criteria:

* Limited mouth opening or symptomatic temporomandibular joint disorder
* Inability to tolerate extended long periodontal treatment and/or hyperactive gag reflex
* Current or former smoker or vape user
* Pregnant and/or breastfeeding
* Having diabetes mellitus type I or II
* Having bleeding disorder or is on anticoagulants
* Underwent periodontal treatment and/or surgery in past 6 months prior
* Undergoing orthodontic therapy, or completed in past 3 months prior
* On or had anti-inflammatory drug(s) in past 3 months prior
* On or had antibiotic(s) in past 3 months prior
* Having autoimmune disorder
* On or had immunosuppressant drug(s) in past 3 months prior
* Undergoing or underwent radio- and/or chemo-therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Periodontal probing depth | Baseline immediately before treatment and 3-months post-operative
  Measurement of periodontal pocket depth from gingival margin to base of pocket using UNC-15 probe with and without research stent
Clinical attachment level | Baseline immediately before treatment and 3-months post-operative
  Sum of measurement of periodontal pocket depth from gingival margin to base of pocket and marginal gingiva level from cementoenamel junction to gingival margin using UNC-15 probe with and without research stent
Number of bleeding sites | Baseline immediately before treatment and 3-months post-operative
  Record of scored, assessed bleeding after periodontal probing

SECONDARY OUTCOMES:
Full mouth plaque score | Baseline immediately before treatment and monthly up to 3-months post-operative
  Record of assessed plaque presence in percentage of all sites and total score using Plaque Index System
Full mouth bleeding score | Baseline immediately before treatment and monthly up to 3-months post-operative
  Record of assessed bleeding on probing in percentage of all sites and total score using modified Sulcular Bleeding Index
Gingival margin level & relative clinical attachment level | Baseline immediately before treatment and 3-months post-operative
  Measurement of marginal gingiva level from cementoenamel junction to gingival margin using UNC-15 probe with and without research stent

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, MAHSA University, Jenjarum, Selangor, Malaysia

REFERENCES:
- [Background] Panda S, Purkayastha A, Mohanty R, Nayak R, Satpathy A, DAS AC, Kumar M, Mohanty G, Panda S, Fabbro MD. Plasma rich in growth factors (PRGF) in non-surgical periodontal therapy: a randomized clinical trial. Braz Oral Res. 2020 Apr 17;34:e034. doi: 10.1590/1807-3107bor-2020.vol34.0034. eCollection 2020. PMID 32321052
- [Background] Loos BG, Needleman I. Endpoints of active periodontal therapy. J Clin Periodontol. 2020 Jul;47 Suppl 22(Suppl 22):61-71. doi: 10.1111/jcpe.13253. PMID 31912527
- [Background] Miron RJ, Horrocks NA, Zhang Y, Horrocks G, Pikos MA, Sculean A. Extending the working properties of liquid platelet-rich fibrin using chemically modified PET tubes and the Bio-Cool device. Clin Oral Investig. 2022 Mar;26(3):2873-2878. doi: 10.1007/s00784-021-04268-x. Epub 2021 Nov 23. PMID 34816309
- [Background] Al-Rihaymee S, Sh Mahmood M. The efficacy of non-surgical platelet-rich fibrin application on clinical periodontal parameters and periostin level in periodontitis: Clinical trial. J Cell Mol Med. 2023 Feb;27(4):529-537. doi: 10.1111/jcmm.17675. Epub 2023 Jan 23. PMID 36691719
- [Background] Narendran N, Anegundi RV, Shenoy SB, Chandran T. Autologous platelet-rich fibrin as an adjunct to non-surgical periodontal therapy-A follow up clinical pilot study. Wound Repair Regen. 2022 Jan;30(1):140-145. doi: 10.1111/wrr.12979. Epub 2021 Oct 22. PMID 34687113
- [Background] Torumtay Cin G, Lektemur Alpan A, Cevik O. Efficacy of injectable platelet-rich fibrin on clinical and biochemical parameters in non-surgical periodontal treatment: a split-mouth randomized controlled trial. Clin Oral Investig. 2023 Dec 28;28(1):46. doi: 10.1007/s00784-023-05447-8. PMID 38153510
- [Background] Shunmuga PD, Tadepalli A, Parthasarathy H, Ponnaiyan D, Cholan PK, Ramachandran L. Clinical evaluation of the combined efficacy of injectable platelet-rich fibrin along with scaling and root planing in the non-surgical periodontal therapy of stage III and grade C periodontitis patients having type 2 diabetes mellitus: A randomized controlled trial. Clin Adv Periodontics. 2024 Sep;14(3):223-231. doi: 10.1002/cap.10266. Epub 2023 Sep 25. PMID 37749861
- [Background] Albonni H, El Abdelah AAAD, Al Hamwi MOMS, Al Hamoui WB, Sawaf H. Clinical effectiveness of a topical subgingival application of injectable platelet-rich fibrin as adjunctive therapy to scaling and root planing: a double-blind, split-mouth, randomized, prospective, comparative controlled trial. Quintessence Int. 2021 Jul 20;52(8):676-685. doi: 10.3290/j.qi.b1492019. PMID 34076375
- [Background] Dohan Ehrenfest DM, Pinto NR, Pereda A, Jimenez P, Corso MD, Kang BS, Nally M, Lanata N, Wang HL, Quirynen M. The impact of the centrifuge characteristics and centrifugation protocols on the cells, growth factors, and fibrin architecture of a leukocyte- and platelet-rich fibrin (L-PRF) clot and membrane. Platelets. 2018 Mar;29(2):171-184. doi: 10.1080/09537104.2017.1293812. Epub 2017 Apr 24. PMID 28437133
- [Background] Kubesch A, Barbeck M, Al-Maawi S, Orlowska A, Booms PF, Sader RA, Miron RJ, Kirkpatrick CJ, Choukroun J, Ghanaati S. A low-speed centrifugation concept leads to cell accumulation and vascularization of solid platelet-rich fibrin: an experimental study in vivo. Platelets. 2019;30(3):329-340. doi: 10.1080/09537104.2018.1445835. Epub 2018 Mar 6. PMID 29509050
- [Background] Wend S, Kubesch A, Orlowska A, Al-Maawi S, Zender N, Dias A, Miron RJ, Sader R, Booms P, Kirkpatrick CJ, Choukroun J, Ghanaati S. Reduction of the relative centrifugal force influences cell number and growth factor release within injectable PRF-based matrices. J Mater Sci Mater Med. 2017 Oct 25;28(12):188. doi: 10.1007/s10856-017-5992-6. PMID 29071440
- [Background] Choukroun J, Ghanaati S. Reduction of relative centrifugation force within injectable platelet-rich-fibrin (PRF) concentrates advances patients' own inflammatory cells, platelets and growth factors: the first introduction to the low speed centrifugation concept. Eur J Trauma Emerg Surg. 2018 Feb;44(1):87-95. doi: 10.1007/s00068-017-0767-9. Epub 2017 Mar 10. PMID 28283682
- [Background] Rodriguez Sanchez F, Verspecht T, Castro AB, Pauwels M, Andres CR, Quirynen M, Teughels W. Antimicrobial Mechanisms of Leucocyte- and Platelet Rich Fibrin Exudate Against Planktonic Porphyromonas gingivalis and Within Multi-Species Biofilm: A Pilot Study. Front Cell Infect Microbiol. 2021 Oct 13;11:722499. doi: 10.3389/fcimb.2021.722499. eCollection 2021. PMID 34722331
- [Background] Castro AB, Herrero ER, Slomka V, Pinto N, Teughels W, Quirynen M. Antimicrobial capacity of Leucocyte-and Platelet Rich Fibrin against periodontal pathogens. Sci Rep. 2019 Jun 3;9(1):8188. doi: 10.1038/s41598-019-44755-6. PMID 31160643
- [Background] Fujioka-Kobayashi M, Miron RJ, Hernandez M, Kandalam U, Zhang Y, Choukroun J. Optimized Platelet-Rich Fibrin With the Low-Speed Concept: Growth Factor Release, Biocompatibility, and Cellular Response. J Periodontol. 2017 Jan;88(1):112-121. doi: 10.1902/jop.2016.160443. Epub 2016 Sep 2. PMID 27587367
- [Background] Miron RJ, Fujioka-Kobayashi M, Sculean A, Zhang Y. Optimization of platelet-rich fibrin. Periodontol 2000. 2024 Feb;94(1):79-91. doi: 10.1111/prd.12521. Epub 2023 Sep 8. PMID 37681522
- [Background] Ghanaati S, Booms P, Orlowska A, Kubesch A, Lorenz J, Rutkowski J, Landes C, Sader R, Kirkpatrick C, Choukroun J. Advanced platelet-rich fibrin: a new concept for cell-based tissue engineering by means of inflammatory cells. J Oral Implantol. 2014 Dec;40(6):679-89. doi: 10.1563/aaid-joi-D-14-00138. PMID 24945603
- [Background] Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, Gogly B. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part I: technological concepts and evolution. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e37-44. doi: 10.1016/j.tripleo.2005.07.008. Epub 2006 Jan 19. PMID 16504849
- [Background] Miron RJ, Gruber R, Farshidfar N, Sculean A, Zhang Y. Ten years of injectable platelet-rich fibrin. Periodontol 2000. 2024 Feb;94(1):92-113. doi: 10.1111/prd.12538. Epub 2023 Nov 30. PMID 38037213
- [Background] Caruana A, Savina D, Macedo JP, Soares SC. From Platelet-Rich Plasma to Advanced Platelet-Rich Fibrin: Biological Achievements and Clinical Advances in Modern Surgery. Eur J Dent. 2019 May;13(2):280-286. doi: 10.1055/s-0039-1696585. Epub 2019 Sep 11. PMID 31509878
- [Background] Herrera D, Sanz M, Kebschull M, Jepsen S, Sculean A, Berglundh T, Papapanou PN, Chapple I, Tonetti MS; EFP Workshop Participants and Methodological Consultant. Treatment of stage IV periodontitis: The EFP S3 level clinical practice guideline. J Clin Periodontol. 2022 Jun;49 Suppl 24:4-71. doi: 10.1111/jcpe.13639. PMID 35688447
- [Background] Sanz M, Herrera D, Kebschull M, Chapple I, Jepsen S, Beglundh T, Sculean A, Tonetti MS; EFP Workshop Participants and Methodological Consultants. Treatment of stage I-III periodontitis-The EFP S3 level clinical practice guideline. J Clin Periodontol. 2020 Jul;47 Suppl 22(Suppl 22):4-60. doi: 10.1111/jcpe.13290. PMID 32383274
- [Background] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S162-S170. doi: 10.1111/jcpe.12946. PMID 29926490
- See also: Process for A-PRF - Videos — https://www.a-prf.com/index.php?option=com_content&view=article&id=138&Itemid=607&lang=en
- See also: Description of S-PRF protocol — https://www.intechopen.com/chapters/84935
- See also: Statement on ASA Physical Status Classification System (2020) — https://www.asahq.org/standards-and-practice-parameters/statement-on-asa-physical-status-classification-system